CLINICAL TRIAL: NCT06026865
Title: Clinical Effect and Molecular Mechanisms of Action of S-adenosylmethionine (SAMe) in Patients With Primary Sclerosing Cholangitis (PSC)
Brief Title: S-adenosylmethionine (SAMe) in Patients With Primary Sclerosing Cholangitis (PSC)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Collaborators: National Science Centre, Poland (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2020/39/O/NZ5/03594
Record Dates: First submitted 2023-06-09; First posted 2023-09-07 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2024-07

CONDITIONS: Primary Sclerosing Cholangitis (PSC)
Keywords: PSC
MeSH Terms: conditions — Cholangitis, Sclerosing | interventions — S-Adenosylmethionine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- S-adenosylmethionine (SAMe) (Experimental): Participants randomized to SAMe Group will receive S-adenosyl-L-methionine 1200 mg/daily (as 2400mg SAMe disulfate tosylate) in tablets in two divided doses (800mg in the morning and 400mg midday) over the period of 6 months. In addition, patients will receive standard treatment with ursodeoxycholic acid (UDCA) at a dose of 13-15 mg/kg b.w.
  Interventions: Dietary Supplement: S-Adenosyl-L-methionine (SAMe)
- Placebo (Placebo Comparator): Patients in Placebo Group will receive a placebo of identical appearance, smell and taste, with the same schedule. In addition, patients will receive standard treatment with ursodeoxycholic acid (UDCA) at a dose of 13-15 mg/kg.In addition, patients will receive standard treatment with ursodeoxycholic acid (UDCA) at a dose of 13-15 mg/kg b.w.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: S-Adenosyl-L-methionine (SAMe) — S-adenosyl-L-methionine 1200 mg/daily as 2400mg S-Adenosyl-L-methionine disulfate tosylate
  Other Names: S-adenosylmethionine
  Arms: S-adenosylmethionine (SAMe)
Other: Placebo — Placebo of identical appearance, smell and taste, with the same schedule.
  Arms: Placebo

SUMMARY:
The aim of this study is to investigate clinical effects (liver biochemistries, health-related quality of life, liver stiffness) and underlying mechanisms of hepatoprotection of S-adenosylmethionine in patients with primary sclerosing cholangitis. The study will be performed in a randomized and placebo-controlled fashion.

DETAILED DESCRIPTION:
The study is designed as a randomised, double-blind, placebo-controlled trial.

Eighty participants will be randomized in 1:1 ratio to one of two arms of the study: Intervention or Placebo. Participants in Intervention Group will be treated with S-adenosyl-L-methionine 1200 mg/daily in tablets in two divided doses (800mg in the morning and 400mg midday) over the period of 6 months. Patients in Placebo Group will receive a placebo of identical appearance, smell and taste, with the same schedule.

Participants will be monitored in out-patient clinic at baseline, interim visits at weeks: 4, 12, end of treatment at 24 weeks and follow-up visit after 4-6 weeks wash-out period. Treatment adherence, adverse events, serum biochemistry and health related quality of life will be assessed at each visit. Liver fibrosis will be measured with transient elastography at baseline and at the end of treatment.

ELIGIBILITY:
Inclusion Criteria:

* primary sclerosing cholangitis fulfilling EASL criteria;
* age: 18 - 75 years;
* treatment with ursodeoxycholic acid (UDCA) in a dose of 13-15mg/kg b.w. for at least 6 months.

Exclusion Criteria:

* inability to give informed consent;
* patients with other forms of chronic liver diseases;
* decompensated liver cirrhosis (Child-Pugh class B-C);
* patients with PSC who underwent stenting of their biliary tree within 6 months;
* other diseases or states that can affect quality of life and mood: decompensated diabetes mellitus, renal insufficiency requiring dialyses, malignancy, heart failure ≥ New York Heart Association (NYHA) II, organ transplantation, known HIV infection, rheumatoid arthritis, asthma, psychiatric disorders;
* treatment with: steroids, statins, rifampicin, antidepressants;
* pregnant or breastfeeding women;
* history of hypersensitivity reactions to S-adenosylmethionine;
* any other condition, which in the opinion of the investigators would impede the patient's participation or compliance in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in liver biochemistries | 6 months
  Change in levels of liver enzymes (Aspartate Transaminase, Alanine Transaminase, Gamma-glutamyltransferase, Alkaline Phosphatase)
Change in Health-related Quality of Life | 6 months
  Change in severity of chronic fatigue and other aspects of health-related quality of life assessed by questionnaire SF-36 (36-Item Short Form Survey).
Change in PSC-related Quality of Life | 6 months
  Change in severity of chronic fatigue and other aspects of health-related quality of life assessed by questionnaire PBC-40.
Change in Quality of Life | 6 months
  Change in severity of generalized anxiety disorder assessed by questionnaire GAD-7 (General Anxiety Disorder-7).
Change in pruritus severity | 6 months
  Change in pruritus severity on the Visual Analogue Scale (VAS) - 0 (no pruritus) to 10 (worst pruritus).
Change in liver stiffness | 6 months
  Change in liver stiffness on liver elastography (measured in kPa)

SECONDARY OUTCOMES:
Molecular assesment of hepatoprotective properties of SAMe | 6 months
  Assessment of changes in antioxidant defence system (assessed as plasma MDA, SOD2, FGF-19, TNF-α, IL6, IL10, TGFβ, INFγ, homocysteine concentrations).

CONTACTS AND LOCATIONS:
Overall Officials: Piotr Milkiewicz, MD, PhD, Principal Investigator — Department of Hepatology, Transplantology and Internal Medicine, Medical University of Warsaw
Locations (1):
- Department of Hepatology, Transplantology and Internal Medicine, Medical University of Warsaw, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No